CLINICAL TRIAL: NCT05675163
Title: Antioxidant and Immune Effects of Vitamin K2 - the ProteK2t Study
Brief Title: Antioxidant and Immune Effects of Vitamin K2
Acronym: ProteK2t
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NIZO Food Research (Other)
Collaborators: Kappa Bioscience AS (Unknown)
Responsible Party: Principal Investigator, Alwine Kardinaal, Principal Scientist Nutrition & Health, NIZO Food Research
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: NL80827.028.22
Record Dates: First submitted 2022-12-22; First posted 2023-01-09 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Oxidative Stress; Inflammation
MeSH Terms: conditions — Inflammation | interventions — Vitamin K 2

STUDY DESIGN:
Intervention Model Description: 3 way crossover trial for evaluating the effect on oxidative stress markers. The first study period, is also used as a parallel study for studying the effect on immune markers.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): matched dose of sunflower oil
  Interventions: Dietary Supplement: Placebo
- Vitamin K2 low dose (Experimental): 333 μg/d Vitamin K2 (MK-7)
  Interventions: Dietary Supplement: Vitamin K2; Dietary Supplement: Placebo
- Vitamin K2 high dose (Experimental): 666 μg/d Vitamin K2 (MK-7)
  Interventions: Dietary Supplement: Vitamin K2

INTERVENTIONS:
Dietary Supplement: Vitamin K2 — (K2VITAL® 1% MCT Oil)
  Arms: Vitamin K2 high dose; Vitamin K2 low dose
Dietary Supplement: Placebo — Sunflower oil
  Arms: Placebo; Vitamin K2 low dose

SUMMARY:
The aim of the study is to obtain insight into a dose-dependent effect of vitamin K2 on oxidative stress and specific markers of the immune system.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported postmenopausal (at least one year after the final menstruation)
* BMI ≥25 and ≤32 kg/m2;
* Plasma dp-ucMGP concentration in highest 50-66% of the screened population
* Non-smoking, defined as not smoking currently and not having smoked (at all) in the year before study start;
* Healthy as assessed by the health questionnaire and according to the judgment of the study physician;
* Voluntary participation;
* Having given written informed consent;
* Willing to comply with study procedures;

Exclusion Criteria:

* Plasma dp-ucMGP concentration >1000 pmol/L at screening
* Treatment with oral antibiotics within 2 months of the start of the study
* Any vaccination in the month before study start or any scheduled vaccination during the study period
* Use of antioxidant or vitamin K and D supplements;
* Use of antioxidant or vitamin K and D supplements in the month before the start of the study;
* Use of aspirin or medication with established antioxidant or anti-inflammatory properties;
* Use of medication that interferes with vitamin K or blood coagulation;
* Use of statins to reduce level of low-density lipoprotein cholesterol in the blood;
* Hyperlipidaemia, diabetes, hypertension, intestinal disease, diseases with an inflammation component;
* Hormone replacement therapy in women;
* Follow a vegetarian or vegan diet;
* Participation in any clinical trial including blood sampling and/or administration of substances up to 30 days before day 1 of this study;
* Alcohol consumption for men > 28 units/week and >4/day; for women: >21 units/week and >3/day;
* Reported unexpected weight loss or weight gain of > 3 kg in the month prior to pre-study screening, or intention to lose weight during the study period;
* Reported slimming or medically prescribed diet;
* Recent blood donation (<1 month prior to Day 01 of the study);
* Not willing to give up blood donation during the study;

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2023-05-16 (Actual); Study Completion 2023-05-16 (Actual)

PRIMARY OUTCOMES:
plasma ox-LDL | 3 weeks
  Dose dependent change in ox-LDL levels

SECONDARY OUTCOMES:
plasma MDA | 3 weeks
  Dose dependent change in plasma MDA levels
plasma CRP | 3 weeks
  Dose dependent change in plasma CRP levels
IL-6 | 3 weeks
  Dose dependent change in plasma IL-6 levels
Phagocytosis capacity | 3 weeks
  % positive and MFI of monocytes and granulocytes
PBMC gene expression | 3 weeks
  Differential Gene Expression analysis (DGE) - Fold change and relative abundance

CONTACTS AND LOCATIONS:
Locations (1):
- NIZO food research, Ede, Netherlands

IPD SHARING:
Plan to Share IPD: No